CLINICAL TRIAL: NCT00439998
Title: Ultrasound Imaging For Facilitating Labour Epidurals in Obese Parturients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 06-03; 06-0218-E
Record Dates: First submitted 2007-02-22; First posted 2007-02-26 (Estimated); Last update posted 2009-07-30 (Estimated); Status verified 2009-07

CONDITIONS: Obesity
Keywords: Ultrasound; Obesity; Needle Depth
MeSH Terms: conditions — Obesity | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Ultrasound — ultrasound scan of the lumbar spine with 2-5 MHz curved array probe

SUMMARY:
The efficacy of an epidural depends mainly on accurate placement of the catheter in the epidural space. Therefore, identification of the epidural space is the most vital part of the procedure. Obese patients represent the most challenging group for the identification of anatomical landmarks. With the use of ultrasound, we can visualize the images of the anatomical structures in the back. Some anesthesiologists believe ultrasound can help in the placement of an epidural, and routinely use it to assist in determining needle entry point in your back as well as estimating the depth at which the epidural space will be found. Our hypothesis is that the use of lumbar spine ultrasound imaging will accurately determine the epidural space depth and the epidural insertion point in obese patients.

DETAILED DESCRIPTION:
Recent technical advances, especially the evolution of ultrasound technology, have helped to some extent in circumventing some of the limitations of epidural anesthesia. The efficacy of an epidural depends mainly on accurate placement of the catheter in the epidural space. Therefore, identification of the epidural space is the most vital part of the procedure. Obese patients represent are the most challenging group for the identification of anatomical landmarks, it is important to determine if ultrasound imaging is a useful technique in this population.

All the patients will undergo ultrasound imaging of the lumbar spine just before epidural insertion. Ultrasound imaging will be performed by one of the investigators. A different anesthesiologist will perform the epidural procedure based on the US information provided by the investigator. The investigator will provide information to the epidural performer on the insertion point, the angle of needle insertion and safe approximate distance before reaching the epidural space to facilitate the epidural performance. To maintain blinding and to prevent performer bias, the exact depth of the epidural space from skin, as seen on the ultrasound will not be disclosed. The investigator, with the aid of an in-built caliper, will measure this distance at a later time before saving the image.

The results of this study are expected to determine the clinical reliability of ultrasound imaging in visualizing the anatomical structures relevant to the technical performance of epidural analgesia in the obese population. Since technical difficulty in performing epidurals is more commonly encountered in obese patients, ultrasound visualization would improve the overall success of the technique by predicting the depth of the epidural needle to be inserted. In turn, the complication rate would be minimized.

ELIGIBILITY:
Inclusion Criteria:

* Full term pregnant patients requesting labor epidurals
* Pre-pregnancy BMI greater than 30

Exclusion Criteria:

* Known spinal deformities
* Previous back instrumentation
* Pre-pregnancy BMI less than 30

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2006-10; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Accuracy of Epidural Depth | 30 minutes

SECONDARY OUTCOMES:
Accuracy of needle angle, re-insertion of the epidural needle in the same interspace or different interspace | 30 minutes
Correlation between BMI and skin thickness | analysis at study end, approximately 1 year
Correlation between BMI and needle depth | analysis at study end, approximately 1 year
Duration of ultrasound scanning | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Mrinalini Balki, MD, Principal Investigator — Department of Anesthesia and Pain Management, Mount Sinai Hospital, University of Toronto
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada